CLINICAL TRIAL: NCT04513912
Title: Double-Blind, Randomized, Parallel-Group Study With Quetiapine Extended Release as Comparator to Evaluate the Efficacy and Safety of Seltorexant 20 mg as Adjunctive Therapy to Antidepressants in Adult and Elderly Patients With Major Depressive Disorder With Insomnia Symptoms Who Have Responded Inadequately to Antidepressant Therapy
Brief Title: A Study of Seltorexant Compared to Quetiapine XR as Adjunctive Therapy to Antidepressants in Adult and Elderly Participants With Major Depressive Disorder With Insomnia Symptoms Who Have Responded Inadequately to Antidepressant Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108810; 42847922MDD3005 (Other: Janssen Research & Development, LLC); 2020-000341-14 (EudraCT Number)
Record Dates: First submitted 2020-08-13; First posted 2020-08-14 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — seltorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Seltorexant (Experimental): Adult participants will receive seltorexant once daily from Day 1-7 and together with matching placebo from Day 8 till Day 182. Elderly participants will receive seltorexant once daily from Day 1-3 and together with matching placebo from Day 4 till Day 182.
  Interventions: Drug: Seltorexant; Drug: Matching placebo to Seltorexant
- Quetiapine Extended-Release (XR) (Active Comparator): Adult participants will receive quetiapine XR once daily from Day 1-2, followed by an increase in dose from Day 3-7, and from Day 8-14 together with matching placebo. After Day 14, quetiapine XR twice daily from Day 14 till Day 182. Elderly participants will receive quetiapine XR once daily from Day 1-3 and twice from Day 4-7, followed by an increase in dose once daily from Day 8-14 together with matching placebo. After Day 14 till Day 182, quetiapine XR will be adjusted by investigator based on the participant's clinical response and tolerability.
  Interventions: Drug: Quetiapine XR; Drug: Matching placebo to Quetiapine XR

INTERVENTIONS:
Drug: Seltorexant — Participants will receive seltorexant over-encapsulated tablet orally.
  Arms: Seltorexant
Drug: Matching placebo to Seltorexant — Participants will receive placebo over-encapsulated tablet matching to seltorexant orally.
  Arms: Seltorexant
Drug: Quetiapine XR — Participants will receive quetiapine XR capsule orally.
  Arms: Quetiapine Extended-Release (XR)
Drug: Matching placebo to Quetiapine XR — Participants will receive placebo capsule matching to quetiapine XR orally.
  Arms: Quetiapine Extended-Release (XR)

SUMMARY:
The purpose of this study is to assess the efficacy of seltorexant compared with quetiapine extended-release (XR) as adjunctive therapy to an antidepressant drug in treatment response in participants with major depressive disorder with insomnia symptoms (MDDIS) who have had an inadequate response to current antidepressant therapy with a selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI).

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a common, serious, recurrent disorder. Seltorexant (JNJ-42847922) is a potent and selective antagonist of the human orexin-2 receptor (OX2R) that is being developed for the adjunctive treatment of MDDIS. The hypothesis for this study is that seltorexant is superior to quetiapine XR in leading to a response after 26 weeks of treatment (greater than or equal to [>=] 50 percent [%] improvement on baseline Montgomery Asberg Depression Rating Scale [MADRS] total score), when administered as adjunctive treatment to an antidepressant in adult and elderly participants with MDDIS who have had an inadequate response to treatment with an SSRI/SNRI. The study will be conducted in 3 phases: a screening phase (up to 30 days), a double-blind (DB) treatment phase (26 weeks), and a post treatment follow-up phase (7 to 14 days after the end of DB treatment phase for all participants, and up to 196 days from baseline for participants who stop study treatment early). The total study duration for each participant will be approximately 32 weeks. Efficacy, safety, pharmacokinetics, and biomarkers will be assessed at specified time points during this study.

ELIGIBILITY:
Inclusion Criteria:

* Meet diagnostic and statistical manual of mental disorders-5th edition (DSM-5) diagnostic criteria for major depressive disorder (MDD), without psychotic features, based upon clinical assessment and confirmed by the structured clinical interview for DSM-5 Axis I disorders-clinical trials version (SCID-CT) diagnosed with first depressive episode prior to age 60. The length of the current depressive episode must be less than or equal to (<=) 24 months
* Have had an inadequate response to at least 1 but no more than 2 antidepressants, administered at an adequate dose and duration in the current episode of depression. The current antidepressant cannot be the first antidepressant treatment for the first lifetime episode of depression. An inadequate response is defined as less than (<) 50 percent (%) reduction but with some improvement (that is, improvement greater than [>] 0%) in depressive symptom severity with residual symptoms present other than insomnia, and overall good tolerability, as assessed by the Massachusetts General Hospital-Antidepressant Treatment Response Questionnaire (MGH-ATRQ)
* Is receiving and tolerating well any one of the following selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) for depressive symptoms at screening, in any formulation and available in the participating country: citalopram, duloxetine, escitalopram, fluvoxamine, fluoxetine, milnacipran, levomilnacipran, paroxetine, sertraline, venlafaxine, desvenlafaxine, vilazodone, or vortioxetine at a stable dose (at or above therapeutic dose level) for at least 6 weeks, and for no greater than 18 months in the current episode
* Have a hamilton depression rating scale (HDRS)-17 total score greater than or equal to (>=) 20 at the first screening interview, must not demonstrate a clinically significant improvement (that is, an improvement of > 20% on their HDRS-17 total score) from the first to the second independent HDRS-17 rating, and must have a HDRS-17 total score >18 at the second screening interview
* Have a patient version insomnia severity index (ISI) total score >= 15 as well as a clinician version of the ISI total score >= 15 at the second screening visit
* Body mass index (BMI) between 18 and 40 kilogram per meter square (kg/m^2), inclusive (BMI=weight/height^2)
* Participant must be medically stable on the basis of the following: physical examination, vital signs (including blood pressure), and 12-lead electrocardiogram (ECG) performed at screening and baseline

Exclusion Criteria:

* Has a recent (last 3 months) history of, or current signs and symptoms of, severe renal insufficiency (creatinine clearance [CrCl] less than [<] 30 milliliter per minute [mL/min]); clinically significant or unstable cardiovascular, respiratory, gastrointestinal, neurologic, hematologic, rheumatologic, immunologic or endocrine disorders. uncontrolled Type 1 or Type 2 diabetes mellitus
* Has a history of treatment-resistant MDD, defined as a lack of response to 2 or more adequate antidepressant treatments in the current episode, as indicated by no or minimal (<25% improvement in symptoms) when treated with an antidepressant of adequate dose (per MGH-ATRQ) and duration (at least 6 weeks)
* Has history or current diagnosis of a psychotic disorder, bipolar disorder, intellectual disability, autism spectrum disorder, borderline personality disorder, somatoform disorders
* Has a history of moderate to severe substance use disorder including alcohol use disorder according to DSM-5 criteria within 6 months before screening
* Has any significant primary sleep disorder, including but not limited to obstructive sleep apnea, restless leg syndrome, or parasomnias. Participants with insomnia disorder are allowed

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 757 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Response (>=50 Percent improvement in MADRS total score from baseline) at Week 26 | Week 26
  Responders are defined as percentage of participants with greater than or equal to (>=) 50 percent (%) improvement in the montgomery-asberg depression rating scale (MADRS) total score from baseline. MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.

SECONDARY OUTCOMES:
Change from baseline in Weight up to Week 26 | Baseline to Week 26
  Change from baseline in weight will be reported.
Time to Study Drug Discontinuation for Potentially Treatment Related Reasons | Up to Week 26
  Time to discontinuation of study drug for potentially treatment related reasons will be reported. Potentially treatment related reasons are defined as all study drug discontinuations excluding the potentially non-treatment related discontinuations (eg, loss of insurance for antidepressant therapy, movement/travel out of the area, change of work-schedule being unable to accommodate visit schedule, family circumstances).
Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score | Baseline to Week 26
  MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The MADRS evaluates the following 10 items: apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Each item is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
Change from Baseline in MADRS-6 Total Score | Baseline to Week 26
  The MADRS-6 scale is a clinician-administered questionnaire used to measure the severity of MDD symptoms. The MADRS-6 scale is a subset of the MADRS-10 scale, comprised of the following individual questionnaire items: Apparent Sadness, Reported Sadness, Inner Tension, Lassitude, Inability to Feel, and Pessimistic Thoughts. Scores range from 0 (no apparent symptoms) to 36 (most severe symptoms).
Change from Baseline in the MADRS Without Sleep Item (MADRS-WOSI) Total Score | Baseline to Week 26
  The MADRS is a 10-item clinician-rated instrument for evaluating severity of symptoms of depression. Each item is rated on a scale from 0 to 6, with higher scores indicating greater symptom severity. MADRS-WOSI considered 9 of the 10 MADRS items, excluding "reduced sleep" item. The total score ranged from 0 to 54, with higher scores corresponding to greater symptom severity.
Change from Baseline in Patient Health Questionnaire, 9-Item (PHQ-9) Total Score | Baseline to Week 26
  The PHQ-9 is a 9-item, participant reported outcome measure to assess depressive symptoms. The scale scores each of the 9 symptom domains of the diagnostic and statistical manual of mental disorders-5th edition (DSM-5) major depressive disorder (MDD) criteria. Each item is rated on a 4 point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms.
Percentage of Participants with Remission (MADRS Total Score less than or equal to (<=) 12) at Week 26 | Week 26
  Percentage of participants with remission (MADRS total Score <=12) will be reported.
Percentage of Participants with a >=50 Percent Improvement in MADRS Total Score and MADRS <=18 at Week 26 | Week 26
  Percentage of participants with a >=50 percent improvement in MADRS total score and MADRS <=18 at Week 26.
Percentage of Participants with Weight Increase >=7 Percent from Baseline at Week 26 | Week 26
  Percentage of participants with weight increase >=7 percent from baseline will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (175):
- United States (75):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - SW Biomedical Research LLC, Tucson, Arizona
  - Proscience Research Group, Culver City, California
  - Pharmacology Research Institute, Encino, California
  - Collaborative NeuroScience Network, Garden Grove, California
  - Collaborative NeuroScience Network, Long Beach, California
  - Pharmacology Research Institute, Los Alamitos, California
  - CalNeuro Research, Los Angeles, California
  - Pharmacology Research Institute, Newport Beach, California
  - NRC Research Institute, Orange, California
  - Pacific Neuropsychiatric Specialists, Orange, California
  - CNRI-Los Angeles, LLC, Pico Rivera, California
  - Prospective Research Innovations Inc, Rancho Cucamonga, California
  - Anderson Clinical Research, Redlands, California
  - University of California at San Diego, San Diego, California
  - National Research Institute, Santa Ana, California
  - CI Trials, Santa Ana, California
  - CMB Clinical Trials, Santee, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Hartford Hospital, Hartford, Connecticut
  - Moonshine Research Center, Inc, Doral, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Indago Research & Health Center Inc, Hialeah, Florida
  - New Life Medical Research Center, Inc., Hialeah, Florida
  - Amedica Research Institute Inc, Hialeah, Florida
  - Meridien Research, Lakeland, Florida
  - Premier Clinical Research, Miami, Florida
  - Global Medical Institutes, Miami, Florida
  - Miami Jewish Health System, Miami, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Synexus Research Orlando, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Compass Research LLC-Bioclinica Research, The Villages, Florida
  - Synexus Clinical Research US Inc, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta LLC, Decatur, Georgia
  - Psych Atlanta, P.C., Marietta, Georgia
  - Chicago Research Center, Chicago, Illinois
  - Capstone Clinical Research, Libertyville, Illinois
  - Alexian Brothers Health System, Lisle, Illinois
  - Baber Research Group, Naperville, Illinois
  - Lemah Creek Clinical Research, Oakbrook Terrace, Illinois
  - Ascension via Christi Research, Wichita, Kansas
  - Riverstar Research, New Orleans, Louisiana
  - Pharmasite Research, Inc., Baltimore, Maryland
  - BTC of New Bedford, New Bedford, Massachusetts
  - Boston Clinical Trials & Medical Research, Roslindale, Massachusetts
  - Psychiatric Care and Research Center (PCRC), O'Fallon, Missouri
  - Bio Behavioral Health, Toms River, New Jersey
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Fieve Clinical Research Inc, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Velocity Clinical Research, Inc., Durham, North Carolina
  - University of Cincinnati, Dept of Psychiatry & Behavioral Neuroscience, Cincinnati, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Neuro Behavioral Clinical Research, North Canton, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, LLC, Oklahoma City, Oklahoma
  - Suburban Research Associates, Pine Hill, Pennsylvania
  - Global Medical Institutes, Scranton, Pennsylvania
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - West Houston Clinical Research Service, Bellaire, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - Hawkins Psychiatry, PC, Mansfield, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Alpine Research Organization, Clinton, Utah
  - Cedar Clinical Research, Draper, Utah
  - University of Virginia, Charlottesville, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Core Clinical Research, Everett, Washington
  - Cary J. Kohlenberg, MD, SC, dba, IPC Research., Waukesha, Wisconsin
- Argentina (11):
  - CENydET - Centro Neurobiologico y de Stress Traumatico, Buenos Aires
  - Hospital Italiano, Buenos Aires
  - FunDaMos, Buenos Aires
  - Hospital Fleni, Ciudad Autonoma Buenos Aires
  - Fundacion Lennox, Córdoba
  - Instituto Privado Kremer, Córdoba
  - Centro Medico Luquez, Córdoba
  - CENPIA, La Plata
  - Clinica Privada de Salud Mental Santa Teresa de Ávila, La Plata
  - CENAIN, Mendoza
  - Clinica Mayo de UMCB, San Miguel de Tucumán
- Belgium (2):
  - AZ Sint-Lucas, Bruges
  - AZ Nikolaas, Sint-Niklaas
- Bulgaria (11):
  - Medical Center Medconsult-Pleven, Pleven
  - MC 'Hipokrat - N', EOOD, Plovdiv
  - Mental Health Center - Rousse, Rousse
  - Medical Center St. Naum, Sofia
  - Medical Center Intermedica, OOD, Sofia
  - MC 'Synexus Sofia' EOOD, Sofia
  - MC 'Synexus Sofia' EOOD, Stara Zagora
  - UMHAT Prof. Dr. St. Kirkovich AD, Stara Zagora
  - State Psychiatric Hospital - Tzarev Brod, Tzarev Brod
  - Diagnostic Consulting Center Mladost - M Varna, Varna
  - Mental Health Center - Veliko Tarnovo EOOD, Veliko Tarnovo
- Canada (3):
  - A.K. Munshi Medical Inc., Sydney, Nova Scotia
  - Canadian Phase Onward, Toronto, Ontario
  - Clinique Force Medic (GCP Trials), Montreal, Quebec
- Czechia (7):
  - Psychiatricka ambulance Saint Anne s.r.o., Brno
  - NeuropsychiatrieHK, s.r.o., Hradec Králové
  - A Shine S R O, Pilsen
  - Clintrial s r o, Prague
  - AD71 s.r.o., Prague
  - NeuropsychiatrieHK, s.r.o., Prague
  - Institut Neuropsychiatricke pece, Prague
- Latvia (4):
  - The Mental Hospital of Jelgava Ģintermuiža - Psychiatry, Jelgava
  - L. Keruze Practice in Psychiatry, Liepāja
  - Hospital of Rezekne, Outpatient Centre of Psychiatry
  - Riga Centre of Psychiatry and Narcology, Riga
- Lithuania (8):
  - Kaunas Silainiu Outpatient Clinic, Public Institution, Kaunas
  - Republic Kaunas Hospital, Kaunas
  - Romuvos Klinika, JSC, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Medical Center Puriena JSC, Šilutė
  - Zirmunai Mental Health Center, Public Institution, Vilnius
  - Antakalnis Psychiatric Consultation Centre, Public Institution, Vilnius
  - Vilnius Mental Health Center, Vilnius
- Malaysia (4):
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Permai, Johor Bahru
  - Hospital Pulau Pinang, Pulau Pinang
  - Hospital Tuanku Jaafar, Seremban
- Poland (10):
  - Gabinet Lekarski Psychiatryczny Ireneusz Kaczorowski, Bełchatów
  - Wlokiennicza MED Specjalistyczna Praktyka Lekarska dr n.med. Tomasz Markowski, Bialystok
  - Przychodnia Srodmiescie SP. z o.o., Bydgoszcz
  - Centrum Badan Klinicznych PI House sp z o o, Gdansk
  - Specjalistyczna Indywidualna Praktyka Lekarska, Lodz
  - CCBR - Lodz - PL, Lodz
  - Specjalistyczna Praktyka Lekarska Marek Domanski, Lublin
  - Synexus Polska Sp. z.o.o. Oddzial w Poznaniu, Poznan
  - Specjalistyczny Osrodek Medycyny Wieku Dojrzalego Sp z o.o., Warsaw
  - Instytut Psychiatrii I Neurologii, Warsaw
- Russia (10):
  - Engels psychiatric hospital, Engel's
  - Kemerovo Regional Clinical Psychiatric Hospital, Kemerovo
  - GUZ Lipetsk Regional psychoneurological Hospital #1, Lipetsk Region
  - JSC Scientific Centre of Personalized Medicine, Moscow
  - FSI Moscow SRI of Psychiatry of Minzdravsocrazvitia, Moscow
  - Moscow Scientific Research Institute of Psychiatry, Moscow
  - Clinical Psychiatry Hospital n.a. N.N. Solodovnikov, Omsk
  - St-Petersburg Bekhterev Psychoneurological Research Institute, Saint Petersburg
  - Klinika StoLet Ltd, Tomsk
  - Sverdlov Regional Psychiatric Clinical Hospital, Yekaterinburg
- Serbia (9):
  - General Hospital Acibadem Bel Medic, Belgrade
  - General Hospital Euromedik, Belgrade
  - Institute of Mental Health Serbia, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - University Clinical Hospital Center Dr Dragisa Misovic- Dedi, Belgrade
  - Special Neuropsychiatric Hospital Kovin, Kovin
  - University Clinical Center Kragujevac, Kragujevac
  - Clinical Center Nis, Niš
  - Specialized Hospital for Neuropsychiatric Diseases Sveti Vracevi, Novi Kneževac
- Slovakia (8):
  - Psychomed-Svatosavsky, s.r.o., Banská Bystrica
  - Nemocnica s poliklinikou Prievidza so sidlom v Bojniciach, Bojnice
  - Epamed sro, Košice
  - Liptovska Nemocnica S Poliklinikou Mudr. Ivana Stodolu, Liptovský Mikuláš
  - Psychiatricka Ambulancia Psycholine S.R.O., Rimavská Sobota
  - FN Trencin, Trenčín
  - Pro mente sana s.r.o., Trenčín
  - Fakultna nemocnica s poliklinikou v Ziline, Žilina
- Ukraine (8):
  - MNCE of Kyiv RC Regional Psychiatric and Narcological Medical Association, Hlevakha
  - Mnpe of Kharkiv Regional Council 'Regional Clinical Psychiatric Hospital #3', Kharkiv
  - Kyiv Territorial Medical Incorporation 'Psychiatry', Kyiv
  - Railway Clinical Hospital #1 of Kiev Railway station of DTGO 'South-Western Railway', Kyiv
  - Medical Center Health and Happy, Kyiv
  - Mnpe 'Regional Clinical Psychiatric Hospital of Kirovohrad Regional Council', Nove
  - Ternopil RCCPH Depts of Psychiatry #2 (m) & Psychiatry #4 (f) Ternopil I.Ya. Gorbachevskyi SMU, Ternopil
  - Zaporizhzhia Regional Clinical Hospital, Zaporizhzhia
- United Kingdom (5):
  - Kingsway Hospital, Derby
  - Synexus, Greater Manchester
  - Garden Valleys Resource Centre, Harrogate
  - Kings College Hospital NHS Trust, London
  - Cornwall Partnership Foundation Trust, Redruth

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson and Johnson is available at www.janssen.com/clinical- trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency